CLINICAL TRIAL: NCT04980313
Title: Effect of a Volumetrically Stable Xenogeneic Collagen Matrix on the Peri-implant Tissues of Immediate Post-extraction Implants: a Randomized Controlled Clinical Study.
Brief Title: Effect of Xenogeneic Collagen Matrix on the Peri-implant Tissues of Immediate Implants.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Octavi Ortiz Puigpelat, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIR-ELC-2021-01
Record Dates: First submitted 2021-06-29; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Xenograft Model
Keywords: immediate dental implants; dental extraction; alveolar socket; connective tissue graft; xenogenic collagen matrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenogenic collagen matrix (Experimental): Volumetrically stable xenogenic collagen matrix
  Interventions: Device: Xenogenic collagen matrix
- Autogenous connective tissue graft (Active Comparator): Autogenous connective tissue graft obtained from the tuberosity area
  Interventions: Device: Autogenous connective tissue graft

INTERVENTIONS:
Device: Xenogenic collagen matrix — Use of xenogenic collagen matrix for the maintenance of buccal soft tissues around immediate dental implantes into extraction sockets.
  Arms: Xenogenic collagen matrix
Device: Autogenous connective tissue graft — Use of connective tissue graft for the maintenance of buccal soft tissues around immediate dental implantes into extraction sockets.
  Arms: Autogenous connective tissue graft

SUMMARY:
The present clinical trial will try to demonstrate the efficacy of stable xenogeneic collagen matrix in maintaining the vestibular coronal soft tissue volume and the stabilization of mid-buccal margin position in immediate post-extraccion sockets compared with the use of autogenous connective tissue grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate oral hygiene (21).
2. Sufficient interocclusal space (≥6 mm) to place a provisional crown without occlusion.
3. Presence of adjacent teeth. Only one tooth gap.
4. Presence of soft tissue and cortical buccal bone of the tooth to be extracted according to the classification of Elian et al. 2007
5. Adequate bone quantity in the apical region of the tooth to be extracted (assessed on the CBCT).

Exclusion Criteria:

1. Patients with medical conditions that affect bone and soft tissue metabolism.
2. Uncontrolled endocrine disorders.
3. Alcohol and drug abuse.
4. Previous history of immunodeficiency syndromes.
5. Patients who smoke> 10 cigarettes a day.
6. Active periodontal disease.
7. Absence of a tooth adjacent to the tooth to be treated.
8. Oral lesions of the untreated mucosa.
9. Recent previous history (<6 months) of local radiotherapy or chemotherapy.
10. Bruxism or severe parafunctions.
11. Pregnant patients.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Analyze the volumetric dimensional changes between the test and the control group | At T0(initial) before extraction
  Analyze the volumetric dimensional changes between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) in mm3.
Analyze the volumetric dimensional changes between the test and the control group | At T6 (6 months after extraction)
  Analyze the volumetric dimensional changes between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) in mm3.
Analyze the volumetric dimensional changes between the test and the control group | At T12 (12 months after extraction).
  Analyze the volumetric dimensional changes between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) in mm3.

SECONDARY OUTCOMES:
Analyze the mid-vestibular gingival level of the treated tooth. | At T0(initial) before extraction
  Analyze the mid-vestibular gingival level of the treated tooth between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) in milimeters.
Analyze the mid-vestibular gingival level of the treated tooth. | At T6 (6 months after extraction)
  Analyze the mid-vestibular gingival level of the treated tooth between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) in milimeters.
Analyze the mid-vestibular gingival level of the treated tooth. | At T12 (12 months after extraction).
  Analyze the mid-vestibular gingival level of the treated tooth between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) with the use of periodontal probe in milimeters.
Measure the band of keratinized tissue around the treated tooth | At T0(initial) before extraction
  Measure the band of keratinized tissue around the treated tooth with the use of a periodontal probe in milimeters.
Measure the band of keratinized tissue around the treated tooth | At T6 (6 months after extraction)
  Measure the band of keratinized tissue around the treated tooth with the use of a periodontal probe in milimeters.
Measure the band of keratinized tissue around the treated tooth | At T12 (12 months after extraction).
  Measure the band of keratinized tissue around the treated tooth with the use of a periodontal probe in milimeters.
Assessment of pain during surgery in both groups | At the day of the surgery
  Assessment of pain during surgery between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) using a numeric scale from 0 to 10, being 0 absence of pain and 10 worst possibble pain.
Assessment of pain during surgery in both groups | After 10 days after surgery
  Assessment of pain during surgery between the test (xenogeneic collagen matrix) and the control group (autogenous connective tissue graft) using a numeric scale from 0 to 10, being 0 absence of pain and 10 worst possibble pain.
Quantification of the analgesic medication intake by patients in both groups | At 10 days after the surgery.
  Quantification of the analgesic medication intake by patients in both groups after 10 days of the surgery. Type of analgesic/antiinflmatory medication and number of pills/day
Comparison of the total surgical time used in each group. | At the day of the surgery
  Measure the time needed for the suergery express in: hh/mm/ss
Comparison of the economic costs for each patient in the collection of the autologous graft and its application versus the purchase of the Fibrogide and its application. | At the day of the surgery
  Comparison of the economic costs for each patient in the collection of the autologous graft and its application versus the purchase of the Fibrogide and its application. Expressed in € per each surgery.
Analyze patient satisfaction between groups | At T0 before extraction.
  Analyze patient satisfaction between groups with the use of a modified Oral Health Impact Profile Questionnaire consisting of 14 questions.
Analyze patient satisfaction between groups | At T12 (12 months after the extraction).
  Analyze patient satisfaction between groups with the use of a modified Oral Health Impact Profile Questionnaire consisting of 14 questions.
Analysis of possible complications in both groups. | They will be reported anytime during the study
  Record the number of complications and also a descriptive analysis of the different types of complications.
Evaluation of implant success in both groups at one year of follow-up | At T12 (12 months after the extraction)
  Evaluation of implant success in both groups at one year of follow-up, expressed in the difference in milimeters of the periimplant bone loss.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dental Ortiz-Puigpelat, Barcelona, Spain